CLINICAL TRIAL: NCT00721409
Title: PHASE 1/2, OPEN-LABEL, RANDOMIZED STUDY OF THE SAFETY, EFFICACY, AND PHARMACOKINETICS OF LETROZOLE PLUS PD 0332991 (ORAL CDK 4/6 INHIBITOR) AND LETROZOLE SINGLE AGENT FOR THE FIRST-LINE TREATMENT OF ER POSITIVE, HER2 NEGATIVE ADVANCED BREAST CANCER IN POSTMENOPAUSAL WOMEN
Brief Title: Study Of Letrozole With Or Without Palbociclib (PD-0332991) For The First-Line Treatment Of Hormone-Receptor Positive Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A5481003; 2008-002392-27 (EudraCT Number)
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: hormone-receptor positive advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): letrozole + PD 0332991
  Interventions: Drug: PD 0332991; Drug: letrozole
- Arm B (Active Comparator): letrozole
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: PD 0332991 — 125 mg/d capsules orally for 3 out of 4 weeks in repeated cycles
  Arms: Arm A
Drug: letrozole — 2.5 mg/d tablets orally on a continuous regimen
  Arms: Arm A
Drug: letrozole — 2.5 mg/d tablets orally on a continuous regimen
  Arms: Arm B

SUMMARY:
The study is aimed to confirm that letrozole + PD 0332991 is safe and tolerable and to assess the effect of the combination on advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Inoperable estrogen receptor positive and HER2 negative breast cancer.
* Postmenopausal status.
* Tumor tissue (archived acceptable) available for biomarker studies. For Phase 2 Part 2 - CCND1 amplification and/or loss of p16 as determined by the central laboratory.
* Acceptable bone marrow, liver and kidney function.

Exclusion Criteria:

* Prior or concomitant treatment for advanced breast cancer.
* Other major cancer in the past 3 years.
* Important cardiovascular events in the past 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 177 (Actual)
Dates: Start 2008-09-15 (Actual); Primary Completion 2013-11-29 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (99):
- United States (46):
  - Central Hematology Oncology Medical group Inc., Alhambra, California
  - UCLA Hematology/Oncology - Alhambra, Alhambra, California
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - UCLA West Medical Pharmacy (Drug Management Only), Los Angeles, California
  - UCLA West Medical Pharmacy, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Drug Management Only: UCLA West Medical Pharmacy, Los Angeles, California
  - Drug Management Only, Los Angeles, California
  - Regulatory Managment, Los Angeles, California
  - TORI -US Central Administration (Regulatory Management), Los Angeles, California
  - TORI -US Central Administration, Los Angeles, California
  - TORI Central Administration (Regulatory Management), Los Angeles, California
  - TORI Central Administration (Regulatory Managment Only), Los Angeles, California
  - TRIO-US Central Administration, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA, Hematology/Oncology, Los Angeles, California
  - Westwood Bowyer Clinic, Peter Morton Medical Building, Los Angeles, California
  - Central Hematology Oncology Medical Group, Inc, Pasadena, California
  - Torrance Health Association, DBA Torrance Memorial Physician Network/Cancer Care Associates, Redondo Beach, California
  - Sansum Santa Barbara Medical Foundation Clinic, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Santa Monica-UCLA Medical Center and Orthopaedic Hospital, Santa Monica, California
  - UCLA Hematology Oncology-Santa Monica, Santa Monica, California
  - UCLA Hematology/Oncology - Santa Clarita, Valencia, California
  - Gwinnett Hospital System Inc.-d/b/a-The Center for Cancer Care, Duluth, Georgia
  - Gwinnett Hospital System Inc.-d/b/a-The Center for Cancer Care, Lawrenceville, Georgia
  - Gwinnett Hospital System Inc.-d/b/a-The Center for Cancer Care, Snellville, Georgia
  - Illinois Cancer Specialists, Chicago, Illinois
  - Resurrection Medical Group, Chicago, Illinois
  - North Shore Oncology-Hematology Associates, Crystal Lake, Illinois
  - North Shore Hematology Oncology, Highland Park, Illinois
  - North Shore Oncology-Hematology Associates, Libertyville, Illinois
  - North Shore Hematology Oncology, Skokie, Illinois
  - Regulatory Office: Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Investigational Products Center (IPC), Fort Worth, Texas
  - US Oncology Research and Clinical Pharmacy, Fort Worth, Texas
  - Virginia Cancer Specialists, PC, Arlington, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
  - Virginia Cancer Specialists, PC, Leesburg, Virginia
  - Virginia Cancer Specialists, PC, Woodbridge, Virginia
- Canada (2):
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - CSSS Champlain-Charles-Le Moyne Local HS-0054, Greenfield Park, Quebec
- France (2):
  - Centre Paul Papin, CRLCC, Angers
  - CHD Vendee, La Roche-sur-Yon
- Germany (11):
  - Gemeinschaftspraxis, Onkologischer Schwerpunkt am Oskar-Helene-Heim, Berlin
  - Gemeinschaftspraxis Haematologie-Onkologie, Dresden
  - Martin-Luther-Universitaet Halle-Wittenberg, Halle
  - Universitaetsklinik und Poliklinik fuer Gynaekologie, Martin-Luther-Universitaet Halle-Wittenberg, Halle
  - Nationales Centrum fuer Tumorerkrankungen, Heidelberg
  - Frauenaerzte Pruener Gang Abts & Partner, Kiel
  - Klinik und Poliklinik fuer Frauenheilkunde und Geburtshilfe Universitaetsklinik Mainz, Mainz
  - Onkolog. Gemeinschaftspraxis, München
  - Frauenklinik vom Roten Kreuz, München
  - Frauenklinik und Poliklinik Klinikum rechts der Isar, Technische Universitaet Muenchen, München
  - Mutterhaus der Borromaeerinnen, Innere Medizin I, Trier
- Hungary (7):
  - Szent Margit Korhaz, Onkologia, Budapest
  - Orszagos Onkologiai Intezet, Kemoterapia B, Budapest
  - Fovarosi Onkormanyzat Uzsoki Utcai Korhaz, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Onkoradiologia, Győr
  - Borsod-Abauj-Zemplen Megyei Korhaz és Egyetemi Oktato Korhaz, Onkologia, Miskolc
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es, Nyíregyháza
  - Markusovszky Egyetemi Oktatokorhaz, Onkoradiologiai Osztaly, Szombathely
- Ireland (5):
  - Bon Secours Hospital, Cork
  - St. Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St. James's Hospital, Dublin
- Italy (7):
  - Divisione Oncologia Medica Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, IRST, Meldola, FC
  - M.O. di Oncologia - Azienda USL di Rimini - Ospedale "Cervesi", Cattolica
  - Ospedale Civile di Faenza Centro Oncologico, Faenza, RA
  - Unita' Operativa di Oncologia, Ospedale Civile di Lugo, Lugo, RA
  - Ospedale Civile di Ravenna, Ravenna
  - Azienda Unita Sanitaria Locale di Rimini, U.O. di Oncologia ed Oncoematologia Ospedale degli Infermi, Rimini
  - Ospedale Villa San Pietro, Roma
- Russia (4):
  - Federal State Budgetary Scientific Institution, Moscow
  - Pyatigorsk Oncology Center, Pyatigorsk
  - State Budgetary Healthcare Institution "Samara Regional Clinical Oncology Dispensary", Samara
  - Republican Clinical Oncology Dispensary of the Ministry of Health of Bashkortostan Republic, Ufa
- South Africa (2):
  - Department of Oncotherapy, National Hospital, Bloemfontein
  - Eastleigh Breast Care Centre, Pretoria
- South Korea (3):
  - National Cancer Center, Center for Breast Cancer, Goyang-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Ico-Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Centro Oncologico de Galicia, A Coruña
  - Hospital General Universitario Vall D'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
- Ukraine (5):
  - Department of Oncology and Medical Radiology, SI "DMA of MOH, Ukraine, "MI "Dnipropetrovsk City, Dnipropetrovsk
  - Municipal Treatment-and-Prophylactic Institution 'Donetsk City Oncological Dispensary' Radiology dep, Donetsk
  - Municipal clinical treatment-and-propyilactic institution "Donetsk regional oncology center',, Donetsk
  - Kyiv City Clinical Oncologic Center, Kyiv
  - Lviv State Oncologic Regional Treatment and Diagnostic Centre, Lviv

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Finn RS, Rugo HS, Gelmon KA, Cristofanilli M, Colleoni M, Loi S, Schnell P, Lu DR, Theall KP, Mori A, Gauthier E, Bananis E, Turner NC, Dieras V. Long-Term Pooled Safety Analysis of Palbociclib in Combination with Endocrine Therapy for Hormone Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: Updated Analysis with up to 5 Years of Follow-Up. Oncologist. 2021 May;26(5):e749-e755. doi: 10.1002/onco.13684. Epub 2021 Mar 10. PMID 33486783
- [Derived] Finn RS, Boer K, Bondarenko I, Patel R, Pinter T, Schmidt M, Shparyk YV, Thummala A, Voitko N, Bananis E, McRoy L, Wilner K, Huang X, Kim S, Slamon DJ, Ettl J. Overall survival results from the randomized phase 2 study of palbociclib in combination with letrozole versus letrozole alone for first-line treatment of ER+/HER2- advanced breast cancer (PALOMA-1, TRIO-18). Breast Cancer Res Treat. 2020 Sep;183(2):419-428. doi: 10.1007/s10549-020-05755-7. Epub 2020 Jul 18. PMID 32683565
- [Derived] Ettl J, Im SA, Ro J, Masuda N, Colleoni M, Schnell P, Bananis E, Lu DR, Cristofanilli M, Rugo HS, Finn RS. Hematologic adverse events following palbociclib dose reduction in patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer: pooled analysis from randomized phase 2 and 3 studies. Breast Cancer Res. 2020 Mar 12;22(1):27. doi: 10.1186/s13058-020-01263-0. PMID 32164785
- [Derived] Rugo HS, Turner NC, Finn RS, Joy AA, Verma S, Harbeck N, Masuda N, Im SA, Huang X, Kim S, Sun W, Iyer S, Schnell P, Bartlett CH, Johnston S. Palbociclib plus endocrine therapy in older women with HR+/HER2- advanced breast cancer: a pooled analysis of randomised PALOMA clinical studies. Eur J Cancer. 2018 Sep;101:123-133. doi: 10.1016/j.ejca.2018.05.017. Epub 2018 Jul 25. PMID 30053671
- [Derived] Dieras V, Rugo HS, Schnell P, Gelmon K, Cristofanilli M, Loi S, Colleoni M, Lu DR, Mori A, Gauthier E, Huang Bartlett C, Slamon DJ, Turner NC, Finn RS. Long-term Pooled Safety Analysis of Palbociclib in Combination With Endocrine Therapy for HR+/HER2- Advanced Breast Cancer. J Natl Cancer Inst. 2019 Apr 1;111(4):419-430. doi: 10.1093/jnci/djy109. PMID 30032196
- [Derived] Wedam SB, Beaver JA, Amiri-Kordestani L, Bloomquist E, Tang S, Goldberg KB, Sridhara R, Ibrahim A, Kim G, Kluetz P, McKee A, Pazdur R. US Food and Drug Administration Pooled Analysis to Assess the Impact of Bone-Only Metastatic Breast Cancer on Clinical Trial Outcomes and Radiographic Assessments. J Clin Oncol. 2018 Apr 20;36(12):1225-1231. doi: 10.1200/JCO.2017.74.6917. Epub 2018 Mar 9. PMID 29522361
- [Derived] Bell T, Crown JP, Lang I, Bhattacharyya H, Zanotti G, Randolph S, Kim S, Huang X, Huang Bartlett C, Finn RS, Slamon D. Impact of palbociclib plus letrozole on pain severity and pain interference with daily activities in patients with estrogen receptor-positive/human epidermal growth factor receptor 2-negative advanced breast cancer as first-line treatment. Curr Med Res Opin. 2016 May;32(5):959-65. doi: 10.1185/03007995.2016.1157060. Epub 2016 Mar 2. PMID 26894413
- [Derived] Finn RS, Crown JP, Lang I, Boer K, Bondarenko IM, Kulyk SO, Ettl J, Patel R, Pinter T, Schmidt M, Shparyk Y, Thummala AR, Voytko NL, Fowst C, Huang X, Kim ST, Randolph S, Slamon DJ. The cyclin-dependent kinase 4/6 inhibitor palbociclib in combination with letrozole versus letrozole alone as first-line treatment of oestrogen receptor-positive, HER2-negative, advanced breast cancer (PALOMA-1/TRIO-18): a randomised phase 2 study. Lancet Oncol. 2015 Jan;16(1):25-35. doi: 10.1016/S1470-2045(14)71159-3. Epub 2014 Dec 16. PMID 25524798
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481003&StudyName=Study%20Of%20Letrozole%20With%20Or%20Without%20Palbociclib%20%28PD-0332991%29%20For%20The%20First-Line%20Treatment%20Of%20Hormone-Receptor%20Positive%20Advanced%20Breast%20Ca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1/2, open-label, randomized study enrolled a total of 12 participants at 3 sites in the United States for Phase 1. Phase 1 participants received Palbociclib + Letrozole. In Phase 2, a total of 165 participants were randomized (84 in palbociclib plus letrozole arm and 81 in letrozole alone arm) at 50 sites in 12 countries.
Pre-assignment Details: Phase 2 portion has 2 parts. Phase 2, Part 1 - ER positive, HER2 negative postmenopausal women with advanced breast cancer. Phase 2, Part 2- ER positive, HER2 negative postmenopausal women with tumors demonstrating CCND1 gene amplification and/or loss of CDKN2A gene.
Groups:
- Phase 1 (Palbociclib + Letrozole): In Cycle 1 (3 weeks), participants received single agent palbociclib 125 mg/d orally for 2 weeks followed by 1 week off treatment. In Cycles 2 and beyond (4 weeks each), participants received letrozole 2.5 mg/d in a continuous regimen plus Palbociclib 125 mg/d orally for 3 weeks followed by 1 week off treatment.
- Phase 2 (Palbociclib + Letrozole): All participants who were randomized to letrozole plus palbociclib in both Phase 2 part 1 (Ph2P1) and Phase 2 part 2 (Ph2P2) are combined and presented. In Ph2P1 and Ph2P2, the participants received palbociclib 125 mg/d orally for 3 weeks followed by 1 week off treatment and letrozole 2.5 mg/d orally in a continuous regimen.
- Phase 2 (Letrozole): All participants who were randomized to receive letrozole alone in both Phase 2 part 1 (Ph2P1) and Phase 2 part 2 (Ph2P2) are combined and presented. This was considered as control arm. Letrozole 2.5 mg/d was administered orally in a continuous regimen.
Period: Overall Study
Arm/Group | Phase 1 (Palbociclib + Letrozole) | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole)
Started | 12 | 84 | 81
Treated | 12 | 83 | 77
Completed | 0 | 2 | 2
Not Completed | 12 | 82 | 79
Not completed — Global deterioration of health status | 2 | 6 | 3
Not completed — Death | 0 | 1 | 0
Not completed — Randomized not Treated | 0 | 1 | 4
Not completed — Reason not specified | 1 | 0 | 2
Not completed — Adverse Event | 0 | 13 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 6 | 5
Not completed — Objective progression or relapse | 8 | 55 | 62

BASELINE CHARACTERISTICS:
Population: Analysis was done on participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 (Palbociclib + Letrozole) | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Total
Number analyzed (Participants) | 12 | 84 | 81 | 177
Age, Customized [Count of Participants; unit: Participants]
  <18 Years | 0 | 0 | 0 | 0
  18-44 Years | 1 | 2 | 4 | 7
  45-64 Years | 6 | 45 | 38 | 89
  >= 65 Years | 5 | 37 | 39 | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 84 | 81 | 177
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 11 | 76 | 72 | 159
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs; All Causalities) at Phase 1
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Maximum treatment duration (approximately 55 months)
Population: Safety analysis set included all participants who received at least 1 dose of any agent of the combination.
Measure: Number; unit: Participants
Arm/Group | Phase 1 (Palbociclib + Letrozole)
Number analyzed (Participants) | 12
Participants
  Participants with AEs | 12
  Participants with SAEs | 2
  Participants with Grade 3 or 4 AEs | 11
  Participants with Grade 5 AEs | 0

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events at Phase 1
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Maximum treatment duration (approximately 55 months)
Population: Safety analysis set included all participants who received at least 1 dose of any agent of the combination.
Measure: Number; unit: Participants
Arm/Group | Phase 1 (Palbociclib + Letrozole)
Number analyzed (Participants) | 12
Participants
  Participants with AEs | 12
  Participants with SAEs | 0
  Participants with Grade 3 or 4 AEs | 11
  Participants with Grade 5 AEs | 0

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities at Phase 1
Description: Dose limiting toxicity was defined as any of the following TEAEs occurring during the second cycle of treatment and possibly attributable to the combination of letrozole plus Palbociclib: 1. Grade 4 hematologic toxicity (including platelets <25,000/μL, ANC <500/μL). 2. Grade 3 neutropenia associated with a documented infection or fever ≥38.5°C. 3. Grade ≥3 non-hematologic toxicities, except those that have not been maximally treated (eg, nausea, vomiting, diarrhea, hypertension). 4. Delay by ≥1 week in receiving the next scheduled dose of either study treatment due to persisting treatment-related toxicities (platelet count <50,000/μL; ANC <1,000/μL; nonhematologic toxicities of Grade ≥3 severity). 5. Inability to deliver at least 80% of the planned Palbociclib or letrozole doses during Cycle 2 due to toxicity possibly attributable to the study treatment.
Time Frame: Cycle 2 (4 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of any agent of the combination.
Measure: Number; unit: Participants
Arm/Group | Phase 1 (Palbociclib + Letrozole)
Number analyzed (Participants) | 12
Participants
  Grade 4 Neutropenia | 2
  <80% of doses due to elevated creatinine | 1

4. Primary Outcome: Progression-Free Survival (PFS) at Phase 2 - Investigator Assessment
Description: PFS was defined as the time from randomization (or the first dose of study treatment for non-randomized studies) to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. PFS calculated as (Weeks or Months) = (first event date minus randomization or the first dose date plus 1) divided by 7 (or 30.44 if in months). PFS is usually characterized by the median, 25% percentile,75% percentile and their 95% Confidence Intervals (CIs).
Time Frame: From randomization date to date of first documentation of progression or death (assessed up to 41 months)
Population: Intent-to-Treat (ITT) was used. This represented all randomized participants from Ph2P1 or Ph2P2 or Ph2P1+Ph2P2, where participants were classified according to the randomized treatment regardless of what treatment, if any, was received.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ph2P1 (Palbociclib + Letrozole): All participants were randomized to receive Letrozole plus Palbociclib. Palbociclib 125 mg/d orally for 3 weeks followed by 1 week off treatment and Letrozole 2.5 mg/d orally in a continuous regimen.
- Ph2P1 (Letrozole): Participants were randomized to receive Letrozole alone. Letrozole 2.5 mg/d was administered orally in a continuous regimen. This was considered as control arm.
- Ph2P2 (Palbociclib + Letrozole): Participants were randomized to receive Letrozole plus Palbociclib. Palbociclib 125 mg/d orally for 3 weeks followed by 1 week off treatment and Letrozole 2.5 mg/d orally in a continuous regimen.
- Ph2P2 (Letrozole): Participants were randomized to receive Letrozole. Letrozole 2.5 mg/d was administered orally in a continuous regimen. This was considered as control arm.
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 84 | 81 | 34 | 32 | 50 | 49
Months | 20.2 [13.8 to 27.5] | 10.2 [5.7 to 12.6] | 26.1 [11.2 to NA] — Not reached | 5.7 [2.6 to 10.5] | 18.1 [13.1 to 27.5] | 11.1 [7.1 to 16.4]
Statistical Analysis 1: Comparison: Phase 2 (Palbociclib + Letrozole) vs Phase 2 (Letrozole); The primary hypothesis to be tested was H0: λ=1 versus. HA: λ<1, where λ was the palbociclib plus letrozole:letrozole alone hazard ratio (HR). A HR less than 1 indicates a reduction in hazard rate in favor of Palbociclib + Letrozole. Stratified analysis was presented above; Test type: Superiority or Other; p = 0.0004, Log Rank — 1-sided p-value from the log-rank test stratified by stratification factors per randomization and Part; Hazard Ratio (HR) = 0.488, 95% CI 2-sided [0.319 to 0.748]
Statistical Analysis 2: Comparison: Ph2P1 (Palbociclib + Letrozole) vs Ph2P1 (Letrozole); The primary hypothesis to be tested was H0: λ=1 versus. HA: λ<1, where λ was the palbociclib plus letrozole:letrozole alone hazard ratio (HR). A HR less than 1 indicates a reduction in hazard rate in favor of Palbociclib + Letrozole. Unstratified analysis was presented above; Test type: Superiority or Other; p < 0.0001, Log Rank — 1-sided p-value from the log-rank test; Hazard Ratio (HR) = 0.299, 95% CI 2-sided [0.156 to 0.572]
Statistical Analysis 3: Comparison: Ph2P2 (Palbociclib + Letrozole) vs Ph2P2 (Letrozole); [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.0046, Log Rank — 1-sided p-value from the log-rank test; Hazard Ratio (HR) = 0.508, 95% CI 2-sided [0.303 to 0.853]

5. Secondary Outcome: Objective Response Rate - Percentage of Participants With Confirmed Objective Tumor Response at Phase 1
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. Per RECIST v1.0: CR defined as disappearance of all target lesions and non-target lesions. PR defined as ≥30% decrease in sum of the longest diameters (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST associated to non-progressive disease response for non target lesions.
Time Frame: From Baseline up to end of study (assessed up to 55 months)
Population: Efficacy analysis set included all enrolled participants with the disease under study, adequate baseline disease assessment, and who started study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1 (Palbociclib + Letrozole)
Number analyzed (Participants) | 12
Percentage of participants | 33.3 [9.9 to 65.1]

6. Secondary Outcome: Percentage of Participants With Clinical Benefit Response (CBR) at Phase 1
Description: CBR is defined as a confirmed CR, confirmed PR, or stable disease (SD) for at least 24 weeks on study according to RECIST. Confirmed responses are those that persisted on repeat imaging >= 4 weeks after initial response.
Time Frame: From Baseline up to end of study (assessed up to 55 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1 (Palbociclib + Letrozole)
Number analyzed (Participants) | 12
Percentage of participants | 83.3 [51.6 to 97.9]

7. Secondary Outcome: Summary of Plasma Palbociclib Steady-state Pharmacokinetic Parameter Following Palbociclib Alone and in Combination With Letrozole: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours (AUC24) at Phase 1
Description: On Cycle 1 Day 14, plasma pharmacokinetic samples were collected prior to and 1, 2, 4, 8, 12, 24, 48, 96 and 120 hours after Palbociclib dosing. On Cycle 2 Day 14, plasma pharmacokinetic samples for Palbociclib and letrozole were collected prior to and 1, 2, 4, 8, 12 and 24 hours after Palbociclib and letrozole dosing.
Time Frame: Cycle 1 Day 14, and Cycle 2 Day 14
Population: The pharmacokinetic concentration set included all participants who were treated and had at least 1 concentration measurement in at least 1 pharmacokinetic assessment day. The pharmacokinetic parameter analysis set consisted of all participants treated who had at least 1 of the pharmacokinetic parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Groups:
- Palbociclib Alone (Cycle 1 Day 14): In Cycle 1 (3 weeks), participants received single agent palbociclib 125 mg/d orally for 2 weeks followed by 1 week off treatment.
- Palbociclib + Letrozole (Cycle 2 Day 14): In Cycles 2 and beyond (4 weeks each), participants received letrozole 2.5 mg/d in a continuous regimen plus palbociclib 125 mg/d orally for 3 weeks followed by 1 week off treatment.
Arm/Group | Palbociclib Alone (Cycle 1 Day 14) | Palbociclib + Letrozole (Cycle 2 Day 14)
Number analyzed (Participants) | 12 | 12
ng·hr/mL | 1982 (29) | 1933 (31)

8. Secondary Outcome: Summary of Plasma Palbociclib Steady-state Pharmacokinetic Parameter Following Palbociclib Alone and in Combination With Letrozole: Maximum Observed Plasma Concentration (Cmax) at Phase 1
Description: as for outcome 7
Time Frame: Cycle 1 Day 14, and Cycle 2 Day 14
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palbociclib Alone (Cycle 1 Day 14) | Palbociclib + Letrozole (Cycle 2 Day 14)
Number analyzed (Participants) | 12 | 12
ng/mL | 115.8 (28) | 108.4 (29)

9. Secondary Outcome: Summary of Plasma Palbociclib Steady-state Pharmacokinetic Parameter Following Palbociclib Alone and in Combination With Letrozole: Time to Maximum Plasma Concentration (Tmax) at Phase 1
Description: as for outcome 7
Time Frame: Cycle 1 Day 14, and Cycle 2 Day 14
Population: as for outcome 7
Measure: Median (Full Range); unit: Hour
Arm/Group | Palbociclib Alone (Cycle 1 Day 14) | Palbociclib + Letrozole (Cycle 2 Day 14)
Number analyzed (Participants) | 12 | 12
Hour | 7.92 (28) [2.17 to 8.20] | 7.92 (29) [2.00 to 8.08]

10. Secondary Outcome: Summary of Plasma Palbociclib Steady-state Pharmacokinetic Parameter Following Palbociclib Alone and in Combination With Letrozole: Terminal Plasma Half-life (t1/2) at Phase 1
Description: as for outcome 7
Time Frame: Cycle 1 Day 14, and Cycle 2 Day 14
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Palbociclib Alone (Cycle 1 Day 14) | Palbociclib + Letrozole (Cycle 2 Day 14)
Number analyzed (Participants) | 12 | 12
Hour | 28.81 (5.0462) [2.17 to 8.20] | NA (NA) [2.00 to 8.08] — Not calculated

11. Secondary Outcome: Summary of Plasma Palbociclib Steady-state Pharmacokinetic Parameter Following Palbociclib Alone and in Combination With Letrozole: Apparent Clearance (CL/F) at Phase 1
Description: as for outcome 7
Time Frame: Cycle 1 Day 14, and Cycle 2 Day 14
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Palbociclib Alone (Cycle 1 Day 14) | Palbociclib + Letrozole (Cycle 2 Day 14)
Number analyzed (Participants) | 12 | 12
L/hr | 63.08 (29) [2.17 to 8.20] | NA (NA) [2.00 to 8.08] — Not calculated

12. Secondary Outcome: Summary of Plasma Palbociclib Steady-state Pharmacokinetic Parameter Following Palbociclib Alone and in Combination With Letrozole: Apparent Volume of Distribution (Vz/F) at Phase 1
Description: as for outcome 7
Time Frame: Cycle 1 Day 14, and Cycle 2 Day 14
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Palbociclib Alone (Cycle 1 Day 14) | Palbociclib + Letrozole (Cycle 2 Day 14)
Number analyzed (Participants) | 12 | 12
L | 2583 (26) [2.17 to 8.20] | NA (NA) [2.00 to 8.08] — Not calculated

13. Secondary Outcome: Summary of Plasma Letrozole Pharmacokinetic Parameter Following Letrozole Alone and in Combination With Palbociclib: AUC24 at Phase 1
Description: On Cycle 2 Day 14, plasma pharmacokinetic samples for Palbociclib and letrozole were collected prior to and 1, 2, 4, 8, 12 and 24 hours after Palbociclib and letrozole dosing. On Cycle 2 Day 28, plasma pharmacokinetic samples were collected prior to and 1, 2, 4, 8, 12, and 24 hours after letrozole dosing.
Time Frame: Cycle 2 Day 14, Cycle 2 Day 28
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·hr/mL
Groups:
- Palbociclib + Letrozole (Cycle 2 Day 14): Participants received 125 mg oral doses of palbociclib with daily 2.5 mg doses of letrozole.
- Letrozole Alone (Cycle 2 Day 28): Participants received daily 2.5 mg doses of letrozole alone.
Arm/Group | Palbociclib + Letrozole (Cycle 2 Day 14) | Letrozole Alone (Cycle 2 Day 28)
Number analyzed (Participants) | 12 | 12
ng·hr/mL | 1739 (30) [2.17 to 8.20] | 1936 (35) [2.00 to 8.08]

14. Secondary Outcome: Summary of Plasma Letrozole Pharmacokinetic Parameter Following Letrozole Alone and in Combination With Palbociclib: Cmax at Phase 1
Description: as for outcome 13
Time Frame: Cycle 2 Day 14, and Cycle 2 Day 28
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palbociclib + Letrozole (Cycle 2 Day 14) | Letrozole Alone (Cycle 2 Day 28)
Number analyzed (Participants) | 12 | 12
ng/mL | 94.95 (27) [2.17 to 8.20] | 104.0 (31) [2.00 to 8.08]

15. Secondary Outcome: Summary of Plasma Letrozole Pharmacokinetic Parameter Following Letrozole Alone and in Combination With Palbociclib: Tmax at Phase 1
Description: as for outcome 13
Time Frame: Cycle 2 Day 14, and Cycle 2 Day 28
Population: as for outcome 7
Measure: Median (Full Range); unit: Hour
Arm/Group | Palbociclib + Letrozole (Cycle 2 Day 14) | Letrozole Alone (Cycle 2 Day 28)
Number analyzed (Participants) | 12 | 12
Hour | 2.00 (27) [0.833 to 4.13] | 1.04 (31) [0.00 to 4.42]

16. Secondary Outcome: Number of Participants With Increase From Baseline in Corrected QT (QTc) Interval at Phase 1
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time corresponding to beginning of depolarization to repolarization of the ventricles (QT interval) was adjusted for RR interval using QT and RR from each ECG by Fridericia's formula (QTcF = QT divided by cube root of RR), by Bazette's formula (QTcB = QT divided by square root of RR) and corrected QT interval according to study-specific criteria (QTcS). Participants with maximum increase from baseline of 30 to less than (<) 60 msec(borderline) and greater than or equal to (>=) 60 msec (prolonged) were summarized.
Time Frame: Cycle 1 Day 1 prior to dosing, Cycle 1 Day 14 (2, 4 [prior to meal], 8, 24, 48, and 96 hours after dosing of Palbociclib), Cycle 2 Day 1 and Day 14 (prior to and 4 hours after dosing of letrozole)
Population: Safety analysis set included all participants who received at least 1 dose of any agent of the combination.
Measure: Number; unit: Participants
Arm/Group | Phase 1 (Palbociclib + Letrozole)
Number analyzed (Participants) | 12
Participants
  QTcB - Change <30 | 9
  QTcB - 30 ≤ change <60 | 3
  QTcB - Change ≥60 | 0
  QTcF - Change <30 | 11
  QTcF - 30 ≤ change <60 | 1
  QTcF - Change ≥60 | 0
  QTcS - Change <30 | 8
  QTcS - 30 ≤ change <60 | 4
  QTcS - Change ≥60 | 0

17. Secondary Outcome: Overall Survival (OS) at Phase 2
Description: Time in weeks or months from randomization to date of death due to any cause. OS was calculated as (the death date or last known alive date (if death date unavailable) minus the date of randomization plus 1) divided by 7 or 30.44 if in months.
Time Frame: From randomization until death (assessed up to 86 months)
Population: ITT was used. This represented all randomized participants from Ph2P1or Ph2P2 or Ph2P1+Ph2P2, where participants were classified according to the randomized treatment regardless of what treatment, if any, was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 84 | 81 | 34 | 32 | 50 | 49
Months | 37.5 [31.4 to 47.8] | 34.5 [27.4 to 42.6] | 37.5 [27.6 to 58.8] | 33.3 [26.0 to 54.3] | 35.1 [28.1 to 47.8] | 35.7 [26.6 to 46.7]
Statistical Analysis 1: Comparison: Phase 2 (Palbociclib + Letrozole) vs Phase 2 (Letrozole); Stratified analysis was presented above. Hazard ratio was assuming proportional hazards, a hazard ratio less than 1 indicated a reduction in hazard rate in favor of palbociclib + letrozole; Test type: Superiority or Other; p = 0.2812, Log Rank — 1-sided p-value from the log-rank test stratified by Part (α = 0.10); Hazard Ratio (HR) = 0.897, 95% CI 2-sided [0.623 to 1.294]
Statistical Analysis 2: Comparison: Ph2P1 (Palbociclib + Letrozole) vs Ph2P1 (Letrozole); Unstratified analysis was presented above; Test type: Superiority or Other; p = 0.2803, Log Rank — 1-sided p-value from the unstratified log-rank test (α=0.10); Hazard Ratio (HR) = 0.837, 95% CI 2-sided [0.458 to 1.527]
Statistical Analysis 3: Comparison: Ph2P2 (Palbociclib + Letrozole) vs Ph2P2 (Letrozole); Unstratified analysis was presented above; Test type: Superiority or Other; p = 0.3875, Log Rank — 1-sided p-value from the unstratified log-rank test (α=0.10); Hazard Ratio (HR) = 0.935, 95% CI 2-sided [0.590 to 1.480]

18. Secondary Outcome: Objective Response Rate - Percentage of Participants With Confirmed Objective Response at Phase 2- Investigator Assessment
Description: Percentage of participants with objective response based assessment of confirmed CR or confirmed PR according to RECIST. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. Per RECIST v1.0: CR defined as disappearance of all target lesions and non-target lesions. PR defined as ≥30% decrease in sum of the longest diameters (LD) of the target lesions taking as a reference the baseline sum LD according to RECIST associated to non-progressive disease response for non target lesions.
Time Frame: From randomization up to the end of treatment (approximately 41 months)
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 84 | 81 | 34 | 32 | 50 | 49
Percentage of participants | 42.9 [32.1 to 54.1] | 33.3 [23.2 to 44.7] | 44.1 [27.2 to 62.1] | 25.0 [11.5 to 43.4] | 42.0 [28.2 to 56.8] | 38.8 [25.2 to 53.8]
Statistical Analysis 1: Comparison: Phase 2 (Palbociclib + Letrozole) vs Phase 2 (Letrozole); Objective Response CI was calculated using the exact Clopper-Pearson method. The stratified analysis presented above was based on CMH test stratified by Part. An Odds Ratio >1 means better response in favor of palbociclib + letrozole arm; Test type: Superiority or Other; p = 0.1347, Cochran-Mantel-Haenszel — 1-sided p-value is from the stratified exact test (1-sided, α =0.10); Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.76 to 2.97]
Statistical Analysis 2: Comparison: Ph2P1 (Palbociclib + Letrozole) vs Ph2P1 (Letrozole); Unstratified analysis was presented above. Exact CI was based on Clopper-Pearson method; Test type: Superiority or Other; p = 0.0849, Chi-squared — Chi-square test was used (1-sided, α=0.10); Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.74 to 7.84]
Statistical Analysis 3: Comparison: Ph2P2 (Palbociclib + Letrozole) vs Ph2P2 (Letrozole); Unstratified analysis was presented above. Exact CI was based on Clopper-Pearson method; Test type: Superiority or Other; p = 0.4515, Chi-squared — Chi-square test was used (1-sided, α=0.10); Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.48 to 2.76]

19. Secondary Outcome: Objective Response Rate - Percentage of Participants With Confirmed Objective Response in Participants With Measurable Disease at Phase 2- Investigator Assessment
Description: Percentage of participants with objective response based assessment of confirmed CR or PR according to RECIST. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. Per RECIST v1.0: CR defined as disappearance of all target lesions and non-target lesions. PR defined as ≥30% decrease in sum of the LD of the target lesions taking as a reference the baseline sum LD according to RECIST associated to non-progressive disease response for non target lesions. Measurable disease referred to the lesions that was accurately measured in at least 1 dimension (longest diameter to be recorded) as ≥20 mm with conventional techniques or as ≥10-16 mm with spiral computer tomography scan (depending on reconstruction interval). Clinical lesions were only be considered measurable when they were superficial (eg, skin nodules, palpable lymph nodes).
Time Frame: From randomization up to the end of treatment (approximately 41 months)
Population: Participants in ITT population with measurable disease were used.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 65 | 66 | 27 | 23 | 21 | 43
Percentage of participants | 55.4 [42.5 to 67.7] | 39.4 [27.6 to 52.2] | 55.6 [35.3 to 74.5] | 34.8 [16.4 to 57.3] | 55.3 [38.3 to 71.4] | 41.9 [27.0 to 57.9]
Statistical Analysis 1: Comparison: Phase 2 (Palbociclib + Letrozole) vs Phase 2 (Letrozole); [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.0471, Cochran-Mantel-Haenszel — 1-sided p-value is from the stratified exact test (1-sided, α =0.10); Odds Ratio (OR) = 1.93, 95% CI 2-sided [0.91 to 4.08]
Statistical Analysis 2: Comparison: Ph2P1 (Palbociclib + Letrozole) vs Ph2P1 (Letrozole); Unstratified analysis was presented above. Exact CI was based on Clopper-Pearson method; Test type: Superiority or Other; p = 0.1180, Chi-squared — Chi-square test was used (1-sided, α=0.10); Odds Ratio (OR) = 2.34, 95% CI 2-sided [0.65 to 8.66]
Statistical Analysis 3: Comparison: Ph2P2 (Palbociclib + Letrozole) vs Ph2P2 (Letrozole); Unstratified analysis was presented above. Exact CI was based on Clopper-Pearson method; Test type: Superiority or Other; p = 0.1631, Chi-squared — Chi-square test was used (1-sided, α=0.10); Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.65 to 4.54]

20. Secondary Outcome: Duration of Response at Phase 2 - Investigator Assessment
Description: Time in weeks, (months or years) from randomization or (start of study treatment for non-randomized studies) to first documentation of objective tumor progression. TTP was calculated as (first event date or last known progression-free date minus the date of randomization [or first dose of study medication for non-randomized studies] plus 1) divided by 7 or 30.44 if in months. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD] per RECIST).
Time Frame: From randomization up to the end of treatment (approximately 41 months)
Population: A subset of ITT population i.e., participants who had response was used for this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 36 | 27 | 15 | 8 | 21 | 19
Months | 20.3 [13.4 to 25.8] | 11.1 [9.3 to 31.6] | 20.9 [6.2 to 25.8] | 10.8 [3.7 to 31.6] | 20.2 [13.0 to NA] — Not reached | 14.8 [7.4 to NA] — Not reached

21. Secondary Outcome: Number of Participants With CBR at Phase 2 - Investigator Assessment
Description: CBR is defined as a confirmed complete response (CR), confirmed partial response (PR), or stable disease (SD) for at least 24 weeks on study according to RECIST.
Time Frame: From randomization up to the end of treatment (approximately 41 months)
Population: ITT was used. This represented all randomized patients from Ph2P1or Ph2P2 or Ph2P1+Ph2P2, where participants were classified according to the randomized treatment regardless of what treatment, if any, was received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 84 | 81 | 34 | 32 | 50 | 49
Percentage of participants | 81.0 [70.9 to 88.7] | 58.0 [46.5 to 68.9] | 76.5 [58.8 to 89.3] | 43.8 [26.4 to 62.3] | 84.0 [70.9 to 92.8] | 67.3 [52.5 to 80.1]
Statistical Analysis 1: Comparison: Phase 2 (Palbociclib + Letrozole) vs Phase 2 (Letrozole); CBR CI was calculated using the exact Clopper-Pearson method. The stratified analysis presented above was based on CMH test stratified by Part. An Odds Ratio >1 means better response in favor of palbociclib + letrozole arm; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel — 1-sided p-value is from the stratified exact test (1-sided, α =0.10); Odds Ratio (OR) = 3.18, 95% CI 2-sided [1.48 to 6.98]
Statistical Analysis 2: Comparison: Ph2P1 (Palbociclib + Letrozole) vs Ph2P1 (Letrozole); Unstratified analysis was presented above. Exact CI was based on Clopper-Pearson method; Test type: Superiority or Other; p = 0.0065, Chi-squared — Chi-square test was used (1-sided, α=0.10); Odds Ratio (OR) = 4.18, 95% CI 2-sided [1.30 to 13.90]
Statistical Analysis 3: Comparison: Ph2P2 (Palbociclib + Letrozole) vs Ph2P2 (Letrozole); Unstratified analysis was presented above. Exact CI was based on Clopper-Pearson method; Test type: Superiority or Other; p = 0.0442, Chi-squared — Chi-square test was used (1-sided, α=0.10); Odds Ratio (OR) = 2.55, 95% CI 2-sided [0.89 to 7.70]

22. Secondary Outcome: Time to Tumor Progression (TTP) at Phase 2-Investigator Assessment
Description: as for outcome 20
Time Frame: From randomization up to the end of treatment (approximately 41 months)
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 84 | 81 | 34 | 32 | 50 | 49
Months | 20.2 [13.8 to 27.5] | 10.2 [5.7 to 12.6] | 26.1 [11.2 to NA] — Not reached | 5.7 [2.6 to 10.5] | 18.8 [13.1 to 27.5] | 11.1 [7.1 to 16.4]
Statistical Analysis 1: Comparison: Phase 2 (Palbociclib + Letrozole) vs Phase 2 (Letrozole); Kaplan-Meier method was applied for median and 95% CI. Hazard ratio was based on assuming proportional hazards, a hazard ratio less than 1 indicates a reduction in hazard rate in favor of palbociclib + letrozole; Test type: Superiority or Other; p < 0.0001, Log Rank — 1-sided p-value is from the stratified log-rank test (α =0.10); Hazard Ratio (HR) = 0.399, 95% CI 2-sided [0.265 to 0.601]
Statistical Analysis 2: Comparison: Ph2P1 (Palbociclib + Letrozole) vs Ph2P1 (Letrozole); Unstratified analysis was presented above. Kaplan-Meier method was applied for median and 95% CI; Test type: Superiority or Other; p < 0.0001, Log Rank — 1-sided p-value is from unstratified log-rank test (α=0.10); Hazard Ratio (HR) = 0.299, 95% CI 2-sided [0.156 to 0.572]
Statistical Analysis 3: Comparison: Ph2P2 (Palbociclib + Letrozole) vs Ph2P2 (Letrozole); Unstratified analysis was presented above. Kaplan-Meier method was applied for median and 95% CI; Test type: Superiority or Other; p = 0.0030, Log Rank — 1-sided p-value is from unstratified log-rank test (α=0.10); Hazard Ratio (HR) = 0.486, 95% CI 2-sided [0.288 to 0.822]

23. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory in Pain Severity Scale (mBPI-sf) Questionnaire at Phase 2
Description: The mBPI-sf is a validated and reliable self-report questionnaire which consists of 13 questions that assess the severity and impact of pain on daily function. The 13 items of the questionnaire make up two scales and two single items. The scales include the 4-item Pain Severity Scale (worst pain, least pain, average pain, and pain right now) and the 7-item Pain Interference Scale (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life). Each item of the pain severity and pain interference scales are based on a 11-point numeric rating scale from 0 ("no pain" or "does not interfere") to 10 ("pain as bad as you can imagine" or "completely interferes").
Time Frame: Baseline, End of treatment (approximately 41 months)
Population: Patient reported outcome evaluable participants included participants who had received at least 1 dose of study medication, had baseline data, and at least one post-baseline measurement.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 76 | 74 | 29 | 27 | 47 | 47
Units on a scale
  Pain at its worst in the last 24 hours | 0.6 (0.42) [28.4 to NA] | 0.1 (0.42) [26.4 to NA] | 0.2 (0.60) [27.6 to NA] | 0.0 (0.89) [26.0 to NA] | 1.2 (0.55) [26.0 to NA] | 0.1 (0.43) [23.4 to NA]
  Pain at its least in the last 24 hours | 0.4 (0.27) | 0.4 (0.27) | 0.3 (0.31) | 0.7 (0.50) | 0.5 (0.40) | 0.2 (0.31)
  Pain on the average | 0.2 (0.33) | 0.2 (0.34) | -0.1 (0.48) | 0.2 (0.64) | 0.4 (0.45) | 0.3 (0.40)
  Pain right now | 0.3 (0.35) | 0.1 (0.36) | 0.1 (0.31) | 0.3 (0.66) | 0.3 (0.55) | 0.0 (0.43)
  Pain Severity Scale | 0.4 (0.29) | 0.2 (0.32) | 0.0 (0.36) | 0.3 (0.62) | 0.6 (0.41) | 0.1 (0.36)
Statistical Analysis 1: Comparison: Phase 2 (Palbociclib + Letrozole) vs Phase 2 (Letrozole); Statistical analysis presented above is for Pain Severity Scale; Test type: Superiority or Other; p = 0.6900, t-test, 2 sided — P-values are based on 2-sample t-test; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.7 to 1.0]
Statistical Analysis 2: Comparison: Ph2P1 (Palbociclib + Letrozole) vs Ph2P1 (Letrozole); Statistical analysis presented above is for Pain Severity Scale; Test type: Superiority or Other; p = 0.7125, t-test, 2 sided — P-values are based on 2-sample t-test; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.8 to 1.2]
Statistical Analysis 3: Comparison: Ph2P2 (Palbociclib + Letrozole) vs Ph2P2 (Letrozole); Statistical analysis presented above is for Pain Severity Scale; Test type: Superiority or Other; p = 0.4012, t-test, 2 sided — P-values are based on 2-sample t-test; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.6 to 1.5]

24. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory in Pain Interference Scale (mBPI-sf) Questionnaire at Phase 2
Description: as for outcome 23
Time Frame: Baseline, End of treatment (approximately 41 months)
Population: as for outcome 23
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 76 | 74 | 29 | 27 | 47 | 47
Units on a scale
  General Activity | 1.1 (0.40) [28.4 to NA] | 0.2 (0.31) [26.4 to NA] | 1.0 (0.66) [27.6 to NA] | 0.2 (0.58) [26.0 to NA] | 1.2 (0.51) [26.0 to NA] | 0.3 (0.37) [23.4 to NA]
  Mood | 0.8 (0.50) | 0.2 (0.36) | 0.6 (0.72) | -0.2 (0.62) | 1.0 (0.69) | 0.4 (0.44)
  Walking ability | 0.8 (0.46) | 0.1 (0.35) | 1.0 (0.55) | 0.3 (0.63) | 0.7 (0.67) | 0.0 (0.43)
  Normal work | 0.7 (0.48) | 0.3 (0.39) | 1.0 (0.53) | 0.2 (0.74) | 0.5 (0.71) | 0.4 (0.45)
  Relations | 0.8 (0.32) | 0.8 (0.32) | 0.6 (0.34) | 0.6 (0.60) | 0.9 (0.47) | 0.8 (0.37)
  Sleep | 0.6 (0.43) | 0.3 (0.35) | 0.1 (0.53) | 0.5 (0.63) | 0.9 (0.61) | 0.1 (0.42)
  Enjoyment of life | 0.8 (0.46) | 0.6 (0.41) | 0.4 (0.34) | 0.2 (0.69) | 1.1 (0.71) | 0.8 (0.52)
  Pain Interference Scale | 0.8 (0.34) | 0.4 (0.30) | 0.7 (0.42) | 0.3 (0.56) | 0.9 (0.48) | 0.4 (0.36)
Statistical Analysis 1: Comparison: Phase 2 (Palbociclib + Letrozole) vs Phase 2 (Letrozole); Statistical analysis presented above is for Pain Interference Scale; Test type: Superiority or Other; p = 0.3346, t-test, 2 sided — P-values are based on 2-sample t-test; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.5 to 1.3]
Statistical Analysis 2: Comparison: Ph2P1 (Palbociclib + Letrozole) vs Ph2P1 (Letrozole); Statistical analysis presented above is for Pain Interference Scale; Test type: Superiority or Other; p = 0.5630, t-test, 2 sided — P-values are based on 2-sample t-test; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.0 to 1.9]
Statistical Analysis 3: Comparison: Ph2P2 (Palbociclib + Letrozole) vs Ph2P2 (Letrozole); Statistical analysis presented above is for Pain Severity Scale; Test type: Superiority or Other; p = 0.4427, t-test, 2 sided — P-values are based on 2-sample t-test; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.7 to 1.6]

25. Secondary Outcome: Presence or Absence of Tumor Tissue Biomarkers at Phase 2 - p16/INK4A, CCND1
Description: Tissue samples were used for retrospective biomarker analyses. For Phase 2 Part 2, the tissue samples were sent to a central laboratory for the assessment of participant selection biomarkers. For Phase 2 Part 1, the assessment of the biomarkers (CCND1 amplification and/or loss of p16) were performed retrospectively from the available samples.
Time Frame: Screening visit (≤ 28 Days prior to dosing)
Population: Copy number analysis set included participants in the Safety Analysis Set who had at least 1 of the biomarker assessments.
Measure: Number; unit: Participants
Arm/Group | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 22 | 24 | 50 | 48
Participants
  CCND1>=1.5 | 12 (0.66) [27.6 to NA] | 9 (0.58) [26.0 to NA] | 39 (0.51) [26.0 to NA] | 44 (0.37) [23.4 to NA]
  p16/INK4A<0.8 | 0 (0.72) | 2 (0.62) | 19 (0.69) | 12 (0.44)
  CCND1>=1.5 and p16/INK4A<0.8 | 0 (0.55) | 2 (0.63) | 8 (0.67) | 8 (0.43)

26. Secondary Outcome: Presence or Absence of Tumor Tissue Biomarkers at Phase 2 - Ki67
Description: Frequency of tumor tissue biomarker Ki67 was evaluated in across treatment groups.
Time Frame: Screening visit (≤ 28 Days prior to dosing)
Population: All participants in the Safety Analysis set who had a Ki67 protein biomarker assessment.
Measure: Number; unit: Participants
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 74 | 71 | 24 | 26 | 50 | 45
Participants
  <=20% | 26 (0.40) [28.4 to NA] | 31 (0.31) [26.4 to NA] | 7 (0.66) [27.6 to NA] | 16 (0.58) [26.0 to NA] | 19 (0.51) [26.0 to NA] | 15 (0.37) [23.4 to NA]
  >20% | 48 (0.50) | 40 (0.36) | 17 (0.72) | 10 (0.62) | 31 (0.69) | 30 (0.44)

27. Secondary Outcome: Presence or Absence of Tumor Tissue Biomarkers at Phase 2 - Tumor Retinoblastoma (RB) and CyclinD1
Description: Presence or absence of tumor RB and CyclinD1 were evaluated. The following definitions of expression applied in the below table: Positive: any expression >0 and Negative: any expression=0.
Time Frame: Screening visit (≤ 28 Days prior to dosing)
Population: Protein biomarkers analysis set included all participants in the safety analysis set who had at least protein biomarker assessment.
Measure: Number; unit: Participants
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 45 | 35 | 12 | 16 | 33 | 19
Participants
  CyclinD1 - Positive | 41 (0.40) [28.4 to NA] | 32 (0.31) [26.4 to NA] | 10 (0.66) [27.6 to NA] | 16 (0.58) [26.0 to NA] | 31 (0.51) [26.0 to NA] | 16 (0.37) [23.4 to NA]
  CyclinD1 - Negative | 3 (0.50) | 3 (0.36) | 2 (0.72) | 0 (0.62) | 1 (0.69) | 3 (0.44)
  RB - Positive | 41 | 32 | 10 | 16 | 31 | 16
  RB - Negative | 2 | 2 | 2 | 0 | 0 | 2

28. Secondary Outcome: Summary of Copy Number for CCND1 (CCND1/CEP11) and p16/INK4A (p16/CEP9) at Phase 2
Description: Gene copy number for CCND1 (CCND1/CEP11) and p16/INK4A (p16/CEP9) were evaluated. This analysis was done for Phase 2 combined group.
Time Frame: Screening visit (≤ 28 Days prior to dosing)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Copy number
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole)
Number analyzed (Participants) | 72 | 72
Copy number
  CCND1 | 2.76 (1.875) [28.4 to NA] | 2.73 (1.559) [26.4 to NA]
  p16/INK4A | 0.83 (0.224) | 0.87 (0.173)

29. Secondary Outcome: Percentage of Participants With Tumor Expression of CYP19A1 and CCND1 Genotypes at Phase 2
Description: One 2-mL blood specimen was collected for the analysis of germline polymorphism in CYP19A1 and CCND1 genes. A single nucleotide polymorphism (SNP) rs4646 as defined in the National Center for Biotechnology Information (NCBI) database in the aromatase gene (CYP19A1) was analyzed. A germline polymorphism G/A870 (rs9344) in the CCND1 gene was analyzed.
Time Frame: Screening visit (≤ 28 Days prior to dosing)
Population: Polymorphism analysis set included participants in the safety analysis set who had at least 1 polymorphism assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 76 | 74 | 30 | 28 | 46 | 46
Percentage of participants
  CYP19A1 - A/A Genotype | 7.9 (0.42) [28.4 to NA] | 5.4 (0.42) [26.4 to NA] | 10.0 (0.60) [27.6 to NA] | 10.7 (0.89) [26.0 to NA] | 6.5 (0.55) [26.0 to NA] | 2.2 (0.43) [23.4 to NA]
  CYP19A1 - C/A Genotype | 34.2 (0.27) | 36.5 (0.27) | 33.3 (0.31) | 42.9 (0.50) | 34.8 (0.40) | 32.6 (0.31)
  CYP19A1 - C/C Genotype | 57.9 (0.33) | 58.1 (0.34) | 56.7 (0.48) | 46.4 (0.64) | 58.7 (0.45) | 65.2 (0.40)
  CCND1 - A/A Genotype | 26.3 (0.35) | 28.4 (0.36) | 33.3 (0.31) | 39.3 (0.66) | 21.7 (0.55) | 21.7 (0.43)
  CCND1 - G/A Genotype | 47.4 (0.29) | 47.3 (0.32) | 43.3 (0.36) | 42.9 (0.62) | 50.0 (0.41) | 50.0 (0.36)
  CCND1 - G/G Genotype | 26.3 | 24.3 | 23.3 | 17.9 | 28.3 | 28.3

30. Secondary Outcome: Number of Participants With TEAEs (All Causalities) at Phase 2
Description: AE:any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship.AEs included both serious and non-serious AEs.SAE:AE resulting in any of following outcomes/deemed significant and jeopardized participants or required treatment to prevent other AE outcomes for any other reason:death;initial or prolonged inpatient hospitalization;life-threatening experience (immediate risk of dying);persistent or significant disability/incapacity;congenital anomaly.Treatment emergent AEs:events occurred between first dose of study drug and up to 28 days after last dose that were absent before treatment or worsened relative to pre-treatment state.AEs were graded as per the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 and coded using Medical Dictionary for Regulatory Activities (MedDRA). Participants with AE of grade 3 or 4 and grade 5 were reported as Grade 3:Severe, Grade 4:Life threatening, Grade 5:Death related to AE.
Time Frame: Baseline up to 28 days after last dose of study drug (for a maximum of 86 months)
Population: All treated as treated set included all treated participants classified by the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 83 | 77 | 33 | 29 | 50 | 48
Participants
  Participants with AEs | 83 | 66 | 33 | 25 | 50 | 41
  Participants with SAEs | 22 | 6 | 10 | 2 | 12 | 4
  Participants with Grade 3 or 4 AEs | 70 | 19 | 29 | 5 | 41 | 14
  Participants with Grade 5 AEs | 1 | 0 | 0 | 0 | 1 | 0

31. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events at Phase 2
Description: AE: any untoward medical occurrence in a participant who received study drug. AEs included both serious and non-serious adverse events. SAE: AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment emergent AEs: events occurred between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. Treatment related AEs: all AEs with causality related to treatment. Relatedness to drug was assessed by the investigator. AEs were graded according to the CTCAE version 3.0 and coded using the MedDRA. Number of participants with AE of grade 3 or 4 and with AE of grade 5 were reported as Grade 3: Severe, Grade 4: Life threatening, Grade 5: Death related to AE.
Time Frame: Baseline up to 28 days after last dose of study drug (for a maximum of 86 months)
Population: All treated as treated set included all treated participants classified by the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
Number analyzed (Participants) | 83 | 77 | 33 | 29 | 50 | 48
Participants
  Participants with AEs | 78 | 33 | 32 | 13 | 46 | 20
  Participants with SAEs | 1 | 0 | 0 | 0 | 1 | 0
  Participants with Grade 3 or 4 AEs | 57 | 2 | 25 | 0 | 32 | 2
  Participants with Grade 5 AEs | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (for a maximum of 86 months)
Description: An event may be categorized as serious in one participant and non serious in another participant, or one participant may experience both serious and non serious event. All treatment emergent AEs and SAEs were collected and reported. The same event may appear as both AE and SAE. All-cause mortality data included all anticipated and unanticipated deaths due to any cause. Analysis was done on participants who received at least one dose of study drug.
Arm/Group | Phase 1 (Palbociclib + Letrozole) | Phase 2 (Palbociclib + Letrozole) | Phase 2 (Letrozole) | Ph2P1 (Palbociclib + Letrozole) | Ph2P1 (Letrozole) | Ph2P2 (Palbociclib + Letrozole) | Ph2P2 (Letrozole)
All-Cause Mortality (participants affected / at risk) | 0/12 | 3/83 | 1/77 | 1/33 | 0/29 | 2/50 | 1/48
Serious Adverse Events (participants affected / at risk) | 2/12 | 22/83 | 6/77 | 10/33 | 2/29 | 12/50 | 4/48
Other Adverse Events (participants affected / at risk) | 12/12 | 83/83 | 57/77 | 33/33 | 22/29 | 50/50 | 35/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 (Palbociclib + Letrozole) (N=12) | Phase 2 (Palbociclib + Letrozole) (N=83) | Phase 2 (Letrozole) (N=77) | Ph2P1 (Palbociclib + Letrozole) (N=33) | Ph2P1 (Letrozole) (N=29) | Ph2P2 (Palbociclib + Letrozole) (N=50) | Ph2P2 (Letrozole) (N=48)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 4 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Palbociclib + Letrozole) (N=12) | Phase 2 (Palbociclib + Letrozole) (N=83) | Phase 2 (Letrozole) (N=77) | Ph2P1 (Palbociclib + Letrozole) (N=33) | Ph2P1 (Letrozole) (N=29) | Ph2P2 (Palbociclib + Letrozole) (N=50) | Ph2P2 (Letrozole) (N=48)
Anaemia (Blood and lymphatic system disorders) | 4 | 29 | 3 | 13 | 0 | 16 | 3
Leukopenia (Blood and lymphatic system disorders) | 8 | 36 | 3 | 16 | 1 | 20 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 2 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 11 | 62 | 4 | 26 | 1 | 36 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 16 | 2 | 8 | 1 | 8 | 1
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 5 | 0 | 2 | 0 | 3 | 0
Lacrimation increased (Eye disorders) | 2 | 3 | 0 | 1 | 0 | 2 | 0
Visual impairment (Eye disorders) | 1 | 4 | 1 | 1 | 1 | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 7 | 4 | 7 | 0 | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 4 | 1 | 1 | 1 | 3
Constipation (Gastrointestinal disorders) | 3 | 13 | 7 | 8 | 4 | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 18 | 9 | 9 | 2 | 9 | 7
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 4 | 2 | 2 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 2 | 1 | 0 | 3 | 2
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 4 | 0 | 0 | 0 | 4 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 25 | 11 | 12 | 7 | 13 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 10 | 2 | 5 | 1 | 5 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 6 | 2 | 1 | 1 | 5 | 1
Vomiting (Gastrointestinal disorders) | 3 | 15 | 3 | 9 | 2 | 6 | 1
Asthenia (General disorders) | 1 | 11 | 4 | 2 | 0 | 9 | 4
Chest pain (General disorders) | 0 | 3 | 4 | 0 | 2 | 3 | 2
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 10 | 34 | 18 | 14 | 7 | 20 | 11
Influenza like illness (General disorders) | 1 | 5 | 2 | 3 | 1 | 2 | 1
Mucosal inflammation (General disorders) | 0 | 7 | 2 | 2 | 0 | 5 | 2
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 6 | 8 | 3 | 5 | 3 | 3
Pain (General disorders) | 2 | 3 | 3 | 1 | 2 | 2 | 1
Pyrexia (General disorders) | 0 | 9 | 2 | 8 | 0 | 1 | 2
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 2 | 1 | 1 | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 3 | 2 | 3 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 3 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 0 | 0
Ear infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 1 | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 1 | 8 | 1 | 4 | 1 | 4 | 0
Localised infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 12 | 7 | 7 | 3 | 5 | 4
Oral herpes (Infections and infestations) | 1 | 3 | 0 | 3 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 0 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 2 | 2 | 1 | 2 | 1 | 0
Skin infection (Infections and infestations) | 2 | 2 | 1 | 2 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 2 | 2 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 12 | 2 | 8 | 2 | 4 | 0
Urinary tract infection (Infections and infestations) | 2 | 9 | 5 | 6 | 3 | 3 | 2
Herpes simplex (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 7 | 3 | 4 | 0 | 3 | 3
Alanine aminotransferase increased (Investigations) | 0 | 6 | 1 | 3 | 1 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 6 | 1 | 2 | 1 | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 8 | 3 | 2 | 2 | 6 | 1
Blood creatinine increased (Investigations) | 2 | 4 | 5 | 1 | 3 | 3 | 2
Blood phosphorus decreased (Investigations) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 4 | 1 | 2 | 0 | 2 | 1
Red blood cell count decreased (Investigations) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 4 | 1 | 0 | 1 | 4 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 17 | 5 | 9 | 2 | 8 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4 | 2 | 2 | 1 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 0 | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 22 | 14 | 9 | 5 | 13 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 17 | 13 | 6 | 5 | 11 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 10 | 3 | 6 | 2 | 4 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3 | 1 | 2 | 4 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 1 | 2 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 9 | 5 | 3 | 3 | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6 | 3 | 2 | 0 | 4 | 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 9 | 7 | 3 | 1 | 6 | 6
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 3 | 1 | 0 | 4 | 3
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 10 | 3 | 3 | 3 | 7 | 0
Dysgeusia (Nervous system disorders) | 1 | 6 | 0 | 4 | 0 | 2 | 0
Headache (Nervous system disorders) | 4 | 12 | 8 | 6 | 3 | 6 | 5
Memory impairment (Nervous system disorders) | 1 | 2 | 1 | 1 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 9 | 4 | 6 | 2 | 3 | 2
Paraesthesia (Nervous system disorders) | 1 | 1 | 2 | 0 | 2 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 4 | 2 | 4 | 0 | 0
Depression (Psychiatric disorders) | 3 | 4 | 5 | 2 | 4 | 2 | 1
Insomnia (Psychiatric disorders) | 3 | 8 | 6 | 4 | 3 | 4 | 3
Mood altered (Psychiatric disorders) | 1 | 4 | 1 | 2 | 0 | 2 | 1
Sleep disorder (Psychiatric disorders) | 0 | 3 | 1 | 0 | 0 | 3 | 1
Dysuria (Renal and urinary disorders) | 3 | 4 | 2 | 2 | 2 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 4 | 1 | 4 | 1 | 0 | 0
Breast discomfort (Reproductive system and breast disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 2 | 4 | 2 | 3 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 2 | 2 | 1 | 0 | 1 | 2
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 12 | 8 | 9 | 4 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 14 | 7 | 4 | 3 | 10 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 1 | 4 | 0 | 5 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 1 | 5 | 0 | 4 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 18 | 2 | 8 | 1 | 10 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 6 | 4 | 2 | 1 | 4 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 1 | 0 | 3 | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 5 | 1 | 3 | 0 | 2 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5 | 2 | 1 | 0 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 7 | 4 | 3 | 1 | 4 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 (0) | 2 | 0 | 2 | 0 | 0 | 0
Hot flush (Vascular disorders) | 3 | 19 | 11 | 9 | 5 | 10 | 6
Hypertension (Vascular disorders) | 0 | 6 | 5 | 1 | 2 | 5 | 3
Lymphoedema (Vascular disorders) | 0 | 4 | 0 | 2 | 0 | 2 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 2 | 1 | 0 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Thyroid mass (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 0
Presbyopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 4 | 2 | 2 | 0 | 2 | 2
Gingivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 0 | 0
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 2 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0
Radicular pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 1 | 0 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 4 | 0 | 2 | 1 | 2
Cellulitis (Infections and infestations) | 0 | 2 | 2 | 2 | 1 | 0 | 1
Weight increased (Investigations) | 0 | 3 | 6 | 1 | 2 | 2 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 0 | 1 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.